CLINICAL TRIAL: NCT01790425
Title: Randomized Controlled Trial Comparing Water vs. Air Method for Performing Colonoscopy in Adult Female Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 319719; UCD IRB # 319719 (Other: UC Davis)
Record Dates: First submitted 2013-01-17; First posted 2013-02-13 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Screening for Colon Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- water colonoscopy (Experimental): The water (study) method: Warm water (body temperature) will be infused into colon to open the lumen for water infusion colonoscopy. Higher rate of complete colonoscopy will be achieved.
  Interventions: Procedure: to infuse water into colon to open the lumen for water infusion colonoscopy
- Air Colonoscopy (Active Comparator): The air (conventional) method: Air is pumped gently (insufflation) into the colon will be used to open the inside space of the colon and aid in colonoscope insertion
  Interventions: Procedure: Air colonoscopy

INTERVENTIONS:
Procedure: to infuse water into colon to open the lumen for water infusion colonoscopy
  Other Names: Water colonoscopy
  Arms: water colonoscopy
Procedure: Air colonoscopy
  Arms: Air Colonoscopy

SUMMARY:
This is a prospective , single center, investigator initiated, randomized controlled trial to compare two methods of performing colonoscopy by experienced colonoscopist. Potential female subjects presenting for colonoscopy at UCD GI Lab will be presented with the study option and will be enrolled if they sign the informed consent.

In recent years, the water infusion method has been reported to have several beneficial effects when studied in veteran patients. These include: significant reduction in discomfort to permit a significantly higher percentage (98% vs. 76%) of veterans to complete scheduled unsedated colonoscopy, lower sedation medication requirement when they accepted the option of minimal pre-medication sedation, more patients completing without sedation (78% vs 54%) when they accepted the on demand sedation and an increase in the yield of adenomas (a type of cancer seen in the colon) in screening and surveillance colonoscopy. Reviewers of the method have repeatedly called for studies using the method in female patients to confirm or refute the findings as most of the veteran patients are male patients.

DETAILED DESCRIPTION:
Study Aim Our aim is to perform a randomized controlled trial comparing air insufflation colonoscopy (conventional method ) vs. water infusion colonoscopy ( study method ) in non veteran female subjects presenting for colonoscopy . Subjects will be randomized 1:1 like the flip of coin.

Study Design This is a prospective, single center, investigator initiated, randomized controlled trial (RCT) to compare the study method (water infusion colonoscopy) with conventional method (air insufflation colonoscopy "pump air to dilate the colon to visualize the colon mucosa) in female patients by experienced colonoscopist. Patients will be classified ASA 1 (No organic, physiologic, biomedical or psychiatric disturbance) and ASA 2 (Mild to moderate systemic diseases which are well controlled including hypertension, diabetes mellitus, asthma, age 70 and over) before colonoscopy procedure.

Research Methods and Procedures The air (conventional) method: Air is pumped gently (insufflation) into the colon will be used to open the inside space of the colon and aid in colonoscope insertion The water (study) method: Warm water (body temperature) will be pumped into the colon in place of air to open the inside of space of the colon and aid in colonoscope insertion After insertion, both methods may use any of the following procedures to advance the colonoscope in to the colon: colonoscope shortening maneuver, abdominal compression, by the assistant, and change of patient position. In both methods air insufflation will be used to distend the colon for inspection, biopsy and polypectomy. Washing of the stool covered mucosa and inspection behind the folds will be performed systematically. After turn around in the rectum, residual air and water will be removed by suction.

Data gathering instruments used in the VA studies will be employed (subject interview questions are attached). Statistical analyses similar to those used in the previous VA studies (Student's t tests, Fischer's exact test, Mann-Whitney U test, etc) will be used to analyze the data.

Biopsy and polypectomy will be performed as usual and all tissues will be submitted for routine histological assessment and the pathology will be recorded.

ELIGIBILITY:
Inclusion Criteria:

-All female patients between the ages of 18 to 80 years scheduled for colonoscopy at UC Davis GI Lab.

Exclusion Criteria:

* Patients who refuse to be randomized to the air or water colonoscopy method.
* Patients who are unable to respond to study questionnaires.
* Patients with partial colon resection

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Cecal intubation | Three years
  Examination of the cecum by endoscopy

SECONDARY OUTCOMES:
Amount of opiate and benzodiazepines used for sedation. | Three years
  The total amount of opiate (either demerol of fentanyl) used for sedation.

OTHER OUTCOMES:
Patient discomfort Patient pain rating during and after procedure | Three years
  Patient's pain score (on a 1-10 scale) during and after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Surinder Mann, M.D., Principal Investigator — UCD
Locations (1):
- University of California, Davis, Sacramento, California, United States